CLINICAL TRIAL: NCT06351254
Title: Effects of Kinesthetic Exercises and Sine Sound Waves on Pain, Range of Motion, Disability and Alignment in Cervical Spondylosis
Brief Title: Kinesthetic Exercises and Sine Sound Waves in Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/01101nayab
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Cervical Spondylosis
Keywords: Alignment, Cervical Spondylosis.
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sine sound waves treatment (Experimental): sine sound waves
  Interventions: Procedure: Sine sound waves
- Kinesthetic exercises (Experimental): Head to neutral head position test and head to target repositioning test
  Interventions: Procedure: Kinesthetic exercises
- Sine sound waves plus kinesthetic exercises (Experimental): Combination of sine sound waves and kinesthetic exercises
  Interventions: Procedure: Sine sound waves plus kinesthetic exercises

INTERVENTIONS:
Procedure: Sine sound waves — Group A 8 participants will be given sine sound waves treatment with the frequency of 80 pulses on C1 vertebrae. Treatment session will be 6 session 3 times a week followed by 6 sessions 2 times a week.
  Other Names: Vibro-percussive waves
  Arms: Sine sound waves treatment
Procedure: Kinesthetic exercises — Kinesthetic exercises was conducted for GROUP 2 8 patients for 6 weeks. Before and after assessment was taken to track patient progress. Cervicocephalic kinesthetic sensibility tests were performed. The first test was Head-to-Neutral Head Position(NHP) repositioning test. In the second repositioning test is Head-toTarget repositioning tests.
  Arms: Kinesthetic exercises
Procedure: Sine sound waves plus kinesthetic exercises — Group C 8 was given combine treatment of sine sound waves and kinesthetic exercises before and after measurement was taken.
  Arms: Sine sound waves plus kinesthetic exercises

SUMMARY:
The goal of this Randomized control trial is to determine the Effect of kinesthetic exercises and sound waves on pain, ROM, shoulder alignment and disability in cervical spondylosis. The main question it aims to answer is:

Weather sine sound and kinesthetic exercise are effective in management of pain, rom, alignment, and disability in patients that are suffering from cervical spondylosis

DETAILED DESCRIPTION:
Cervical spondylosis is a progressive disease defined by degenerative changes affecting the vertebrae, intervertebral disks, facets, and associated ligaments. Symptoms of cervical spondylosis manifest as neck pain and neck stiffness and can be accompanied by radicular symptoms when there is compression of neural structures. The degenerative changes are intervertebral disc degeneration, osteophyte formation, and ligamentum flavum and facet hypertrophy. The sine sound waves approach aims to provide orthopaedic spinal treatment through focused vibroacoustic treatment (fVAT) and manage the biomechanical aspect of back pain. Vibroacoustic therapy has been indicated for patients with a range of musculoskeletal, neurological, and haemodynamic problems demonstrating positive changes in pain, spasticity, movement control, and specifically fatigue and anxiety in those with spinalcord or brain injuries. For neck pain syndromes, the kinesthetic rehabilitation exercises (i. e.,eye-follow exercises, head relocation exercises, eye-head coordination, and gaze stability exercises) are developed to improve or restore somatosensory and sensorimotor function by enhancing tactile afferents cues. Kinaesthetic exercises have an added advantage over the conventional exercise programs as it uses an unconscious component of proprioceptive signals for the automatic control of cervical muscle tone and posture.

The research include 3 intervention groups Group A will be give sine sound waves treatment 6 sessions 3 times a week followed by 6 sessions 2 times a week. Group B will be given kinesthetic exercise for 6 weeks. And group C will be given combination of both group A and group B treatments. Outcomes, encompassing pain levels, range of motion (ROM), and Neck Disability Index (NDI) scores, will be evaluated using the Numeric Pain Rating Scale, Goniometer, and Crom device. Data analysis will employ SPSS version 26. Data will be collected at baseline, immediately post-intervention, and at follow-up intervals. Statistical analyses will be conducted to assess and compare the effects of the interventions on the primary and secondary outcomes, thereby addressing the research question regarding their relative efficacy.

ELIGIBILITY:
Inclusion Criteria:

* neck pain
* age 45-60 years
* radiography showed degenerative changes

Exclusion Criteria:

* cervical myelopathy
* whiplash injury
* infection involving the c-spine

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
NPRS | 6 weeks
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Inclinometer | 6 weeks
  An inclinometer (or clinometer), is an instrument used for measuring the angles of slope/tilt and elevation/depression of an object with respect to gravity. The resulting measurement is either given an angular measurement (degrees, minutes, seconds etc.) or as a percentage with reference to a level zero plane.
Goniometer | 6 weeks
  A goniometer is the most common instrument used to measure range of motion. If a patient has altered range of motion in a particular joint, the therapist can use a goniometer to assess what the range of motion is at the initial assessment, and then make sure the intervention is working by using the goniometer in subsequent sessions to assess the effectiveness of the intervention.
NDI | 6 weeks
  Patient neck disability index is assessed through this index

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, Ms, Principal Investigator — Riphah
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No